CLINICAL TRIAL: NCT01310283
Title: Caries Management by Risk Assessment in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ling Zhan, Asisstant professor in residence, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A106017
Record Dates: First submitted 2011-03-04; First posted 2011-03-08 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Dental Caries
Keywords: dental caries; children; mutans streptococci; lactobacilli; cariogenic bacteria
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- control group (No Intervention): Conventional pediatric dental care.
  Interventions: Other: xylitol mints and fluoride varnish

INTERVENTIONS:
Other: xylitol mints and fluoride varnish — Subjects in the intervention group will receive additional diet, oral hygiene handouts, more frequent professional fluoride application, and xylitol mints based on their caries risk levels.

SUMMARY:
The goal of this study is to address the effectiveness of a modified cavity prevention protocol for 5-9 year-old children which emphasizes better diet modification, more frequent professional fluoride applications, and xylitol product usage based on individual risk status in a 1-year randomized controlled clinical trial in the University of California, San Francisco (UCSF) Tenderloin Community Pediatric Dental Clinic. The investigators hypothesize that the regimen will help to reduce new cavities in children who are at risk for dental cavities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of record at the UCSF Pediatric Dental Clinic, or the UCSF Tenderloin Community Pediatric Dental Clinic, and must be:
2. Patients of record at the Tenderloin community and UCSF pediatric dental clinics
3. 5-9 years old

3. Be able to give informed assent, consent and answer questionnaires in English, Spanish or Chinese by parents or guardian 4. Be unlikely to move from the area during the study period 5. Be willing to participate regardless of group assignment and comply with all study procedures

Exclusion Criteria:

Persons with:

1. Prolonged antibiotic use in the past three months.
2. Dental needs outside of the community pediatric clinics, such as care provided in specialty clinics

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
new decayed surfaces | 1 year

SECONDARY OUTCOMES:
cariogenic bacteria levels | 6 month and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zhan, DDS, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Pediatric Dental Clinic at UCSF, School of Dentistry and UCSF Pediatric Dentistry Clinica at the Tenderloin Community School, San Francisco, California
  - The Pediatric Dentistry Clinic at UCSF and Tenderloin Community Elementary School, San Francisco, California